CLINICAL TRIAL: NCT04030052
Title: Emicizumab PUPs and Nuwiq ITI Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The Emi PUPs and Nuwiq ITI study has been closed due to slow enrollment and study site startup.
Sponsor: Emory University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Sidonio, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00111805
Record Dates: First submitted 2019-07-21; First posted 2019-07-23 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hemophilia A
Keywords: safety; immunogenicity; hemostatic efficacy; prophylactic; infants; children; hemostasis; hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; Clinical Protocols; simoctocog alfa (Nuwiq); emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Untreated/minimally treated moderate HA no inhibitors (Experimental): Previously untreated patients (PUPs) and minimally treated patients (MTPs) <3 years of age with moderately severe (≤2% FVIII) HA and no inhibitors.
  Interventions: Drug: Nuwiq (low dose protocol); Drug: HEMLIBRA
- Treated any moderate HA with existing inhibitors (Experimental): Children <21 years of age with moderately severe (≤2% FVIII) HA and with already existing inhibitors (LTI or HTI).
  Interventions: Drug: HEMLIBRA; Drug: Nuwiq (Atlanta protocol)

INTERVENTIONS:
Drug: Nuwiq (low dose protocol) — After receiving HEMLIBRA® for 1-6 months, rFVIII (NUWIQ®) will be given at low dose (25 ±5 units/kg/dose) every 7-14 days as part of a low dose factor exposure program and for on demand use for acute bleeding episodes/procedures. NUWIQ® will be administered intravenously (IV) via peripheral infusion. If the infant has a central line such as a PICC line or mediport this can be used.
  Other Names: Simoctocog alfa
  Arms: Untreated/minimally treated moderate HA no inhibitors
Drug: HEMLIBRA — Four weekly subcutaneous (SQ) injections of HEMLIBRA® loading doses of 3 mg/kg will be given. A total of 12 mg/kg within the first month is allowed for the loading doses. Maintenance dosing will follow, and will either be 1.5 mg/kg/dose weekly, 3 mg/kg/dose biweekly (every 2 weeks), or 6 mg/kg/dose every 4 weeks depending on the recommended dosing.
  Other Names: Emicizumab, ACE910, and RO5534262
Drug: Nuwiq (Atlanta protocol) — After completing HEMLIBRA® loading doses, participants will receive intravenous (IV) infusions of NUWIQ® 3 times per week, 100 units/kg the Atlanta protocol. Infusions will be given at least 36 hours from the previous NUWIQ® injection. Participants will continue on the HEMLIBRA® SQ - NUWIQ® IV treatment regimen for up to 12 months of NUWIQ® treatment.
  Other Names: Simoctocog alfa
  Arms: Treated any moderate HA with existing inhibitors

SUMMARY:
This study prospectively investigates the safety, FVIII immunogenicity, and hemostatic efficacy of prophylactic HEMLIBRA® given with a concomitant low dose recombinant factor VIII (rFVIII) known as NUWIQ®, in HA infants and children <3 years old who have had little to no previous exposure to FVIII. In addition, the study investigates the safety and efficacy of a novel FVIII ITI regimen in children <21 with existing low and high titer inhibitors (LTI and HTI).

DETAILED DESCRIPTION:
Hemophilia A (HA) is a congenital bleeding disorder caused by deficient or dysfunctional factor VIII (FVIII) which leads to bleeding correlated with severity. Management is focused on FVIII replacement in reaction to a bleed or preventive as prophylaxis. Effective treatment is complicated by the: (1) difficulty to administer standard replacement therapy via intravenous injection especially in infants and young children; and (2) development of inhibitors (FVIII neutralizing antibodies). Inhibitors can increase morbidity and mortality and exponentially raise the cost of health care. Although inherited and environmental risk factors for inhibitor formation have been identified, there is no effective strategy to prevent inhibitors from developing. Emicizumab (HEMLIBRA®) was recently approved by the Food and Drug Administration (FDA) in infants, children, and adults with congenital hemophilia A, with and without inhibitors, and offers hemostatic efficacy while reducing the burden of administration since it is given weekly, biweekly (every 2 weeks), or monthly via subcutaneous (SQ) route compared to the intravenous (IV) route of FVIII.

This study prospectively investigates the safety, FVIII immunogenicity, and hemostatic efficacy of prophylactic HEMLIBRA® given with a concomitant low dose recombinant factor VIII (rFVIII) known as NUWIQ®, in HA infants and children <3 years old who have had little to no previous exposure to FVIII. In addition, the study investigates the safety and efficacy of a novel FVIII ITI regimen in children <21 with existing low and high titer inhibitors (LTI and HTI).

ELIGIBILITY:
Inclusion Criteria - Part A:

* Moderately severe (≤2% FVIII) hemophilia A
* <3 Years of age at the time of informed consent
* Caregiver (parent or legal guardian) has provided written informed consent
* ≤2 EDs to pdFVIII, rFVIII, or a single dose of FFP, Cryoprecipitate or PRBCs.
* Adequate hematologic function (HgB >8 g/dL and platelet count >100,000 µL)
* Adequate hepatic function (total bilirubin ≤1.5x ULN and both AST/ALT ≤3x ULN at screening (excluding known Gilbert's)
* Adequate renal function (≤2.5 x ULN and CrCl ≥30 mL/min)
* Negative test for inhibitor (<0.6 BU/mL) with a 72-hour washout within 4 weeks of enrollment
* No documented FVIII inhibitor since birth *Participants will be encouraged to co-enroll in the ATHN 8 Study

Inclusion Criteria - Part B

* Moderately severe (≤2% FVIII) hemophilia A
* <21 Years of age at the time of informed consent
* Documented on 2 occasions a persistent low (>0.6 BU/mL) titer inhibitor with a 72-hour washout within 24 weeks of enrollment or historical high titer inhibitor (>5 BU/mL) and a single occasion of a low titer inhibitor (>0.6 BU/mL) with a 72-hour washout within 24 weeks of enrollment after either the first time ITI or after single attempt of <6 months of continuous 3x/week factor ITI
* Has completed loading doses of HEMLIBRA® (weekly for 4 weeks, dose 3 mg/kg, a total of 12 mg/kg/dose will also be allowed)
* Caregiver and/or participant provided written informed consent
* Adequate hematologic function (HgB >8 g/dL and platelet count >100,000 µL)
* Adequate hepatic function (total bilirubin ≤1.5x ULN and both AST/ALT ≤3x ULN at screening (excluding known Gilbert's)
* Adequate renal function (≤2.5 x ULN and CrCl ≥30 mL/min)

Exclusion Criteria - Part A and B

* Inherited or acquired bleeding disorder other than severe hemophilia A (participants with previous documentation of low von Willebrand factor (vWF) defined as vWF antigen and vWF ristocetin cofactor both between 40-50 will be permitted)
* Previous or current treatment for thromboembolic disease or signs of thromboembolic disease
* Conditions that may increase the risk of bleeding or thrombosis. Will not require or request a thrombophilia evaluation
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the HEMLIBRA® injection (with the exception of rituximab)
* Known HIV infection with CD4 count <200 cells/µL within 24 weeks prior to screening. Testing is not required if can demonstrate negative testing in the mother prior to pregnancy
* Use of systemic immunomodulators at enrollment or planned use during the study
* Participants who are at high risk for thrombotic microangiopathy (TMA) (for example, have a previous medical or family history of TMA), in the investigator's judgment
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose an additional risk, or would, in the opinion of the investigator, preclude the participant's safe participation in and completion of the study
* Planned surgery (excluding minor procedures or central line placement) during the study
* Receipt of HEMLIBRA® as part of a prior investigational study; an investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of the last drug administration; a non-hemophilia-related investigational drug concurrently, within the last 30 days or 5 half-lives, whichever is shorter

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of inhibitors to FVIII | Duration of the follow up (up to 36 months)
  Cumulative incidence of inhibitors to FVIII will be recorded
Number of Immune Tolerance Induction (ITI) success cases | Duration of the follow up (up to 36 months)
  ITI success case is confirmed if three of below are criteria met:
  1. Inhibitor titre < 0.6 BU/mL for at least 2 consecutive measurements
  2. FVIII recovery ≥ 66% of the predefined reference value of 1.5% IU/kg BW approximately 15 to 30 min post-injection
  3. Half-life of FVIII ≥ 6 h
Number of Immune Tolerance Induction (ITI) partial success cases | Duration of the follow up (up to 36 months)
  ITI partial success case is confirmed if two of below criteria are met:
  1. Inhibitor titre < 0.6 BU/mL for at least 2 consecutive measurements
  2. FVIII recovery ≥ 66% of the predefined reference value of 1.5% IU/kg BW approximately 15 to 30 min post-injection
  3. Half-life of FVIII ≥ 6 h
Number of Immune Tolerance Induction (ITI) partial response cases | Duration of the follow up (up to 36 months)
  ITI partial response case is confirmed if one of below criteria is met:
  1. Inhibitor titre < 0.6 BU/mL for at least 2 consecutive measurements
  2. FVIII recovery ≥ 66% of the predefined reference value of 1.5% IU/kg BW approximately 15 to 30 min post-injection
  3. Half-life of FVIII ≥ 6 h
Number of Immune Tolerance Induction (ITI) partial failure cases | Duration of the follow up (up to 36 months)
  ITI partial failure case is confirmed if none of below criteria are met, but participant who initially had a high-titre inhibitor (≥ 5 BU/mL) has a low-titre inhibitor (< 5 BU/mL) at end of ITI.
  1. Inhibitor titre < 0.6 BU/mL for at least 2 consecutive measurements
  2. FVIII recovery ≥ 66% of the predefined reference value of 1.5% IU/kg BW approximately 15 to 30 min post-injection
  3. Half-life of FVIII ≥ 6 h
Number of Immune Tolerance Induction (ITI) failure cases | Duration of the follow up (up to 36 months)
  ITI failure case is confirmed if none of below criteria are met:
  1. Inhibitor titre < 0.6 BU/mL for at least 2 consecutive measurements
  2. FVIII recovery ≥ 66% of the predefined reference value of 1.5% IU/kg BW approximately 15 to 30 min post-injection
  3. Half-life of FVIII ≥ 6 h

SECONDARY OUTCOMES:
Number of joint bleeding events over time (≥3 bleeds in the same joint over the last 24 weeks) | 6 months follow up
  Number of joint bleeding events over time (≥3 bleeds in the same joint over the last 24 weeks) will be recorded
Number of target joint bleeding events over time (≥3 bleeds in the same joint over the last 24 weeks) | 12 months follow up
  Number of target joint bleeding events over time (≥3 bleeds in the same joint over the last 24 weeks) will be recorded
Annualized bleeding rate (ABR) | Duration of the follow up (up to 36 months)
  Number of bleeding events over time (bleed rate) will be recorded to calculate ABR to determine hemostatic efficacy of treatment regiments. Annualized bleeding rate (bleeds/year) is calculated as the number of bleeding events divided by length of time of the treatment regimen.
Number of adverse events | Duration of the follow up (up to 36 months)
  Number of adverse events (AEs and SAEs) will be recorded to evaluate safety of treatment regiments
Change in blood levels of anti-FVIII antibodies | Weekly x4 (±3 days), then monthly (±7 days) up to 36 months
  Blood test will be done to evaluate blood levels of anti-FVIII antibodies
Change in blood levels of anti-Emicizumab antibodies | Weekly x4 (±3 days), then monthly (±7 days) up to 36 months
  Blood test will be done to evaluate blood levels of anti-Emicizumab antibodies
Number of infusions of Nuwiq/Novo7 for treatment of an acute bleeding episode | Duration of the follow up (up to 36 months)
  Number of infusions of Nuwiq/Novo7 for treatment of an acute bleeding episode will be recorded
Number of infusions of rFVIII or rFVIIa for treatment of an acute bleeding episode | Duration of the follow up (up to 36 months)
  Number of infusions of rFVIII or rFVIIa for treatment of an acute bleeding episode will be recorded
Change in blood levels of emicizumab (HEMLIBRA®) in young children (1 month to 24 months of age) | Weekly for 4 weeks, monthly for 5 months, and every 3 months until study end (up to 36 months)
  Blood levels of emicizumab (HEMLIBRA®) in young children (1 month to 24 months of age) will be measured to study Emicizumab pharmacokinetics
Microbiota composition of stool in infants with vs. without inhibitors | Duration of the follow up (up to 36 months)
  Microbiota composition of stool in infants with vs. without inhibitors will be measured
Change in CATCH scale score | Baseline, 36 months
  Scores are calculated as the mean of scores for all items, if 50% or more of the items are missing, then the score is set at missing.
  CATCH scores range from 0 to 100, with the following interpretation:
  * Higher score = Higher the perceived risk to have a bleed while doing daily activities
  * Higher score = Higher impact of hemophilia on daily activities
  * Higher score = Higher the perceived risk to have a bleed while doing social activities
  * Higher score = Higher impact of hemophilia on social activities
  * Higher score = Higher the perceived risk to have a bleed while doing recreational activities
  * Higher score = Higher impact of hemophilia on recreational activities
  * Higher score = Higher impact of hemophilia on work/school activities
  * Higher score = Greater preoccupation related to hemophilia
  * Higher score = Greater perceived burden of the hemophilia treatment
Change in Adapted Inhib-QoL scale score | Baseline, 36 months
  Adapted Inhib-QoL scores range from 0 to 100, with lower scores reflecting better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sidonio, MD, Principal Investigator — Emory University
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Emory University/Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Mindy_L_Simpson@rush.edu, Indianapolis, Indiana
  - Children's Hospital of Michigan/ Wayne State University, Detroit, Michigan
  - Weill Cornell Medicine, New York, New York
  - University of North Carolina - Hemophilia and Thrombosis Center, Chapel Hill, North Carolina
  - Verisiti, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures and appendices) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available beginning 9 months and ending 36 months after publication
Access Criteria: Data will be shared with investigators/researchers involved in the study approved by the steering committee following verification of sound science for the purpose of achieving aims of the study, meta-analysis and for sound scientific evaluation deemed by the steering committee. Proposal may be submitted up to 36 months following publication and can be accessed following steering committee approval directed to Traci Leong (tleong@emory.edu), the statistician.